CLINICAL TRIAL: NCT07222618
Title: "Selfie" Videos: A Novel, Patient-centered, Comprehensive Approach to Measuring Function in MS
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 21-33227
Record Dates: First submitted 2025-10-27; First posted 2025-10-30 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis (MS) - Relapsing-remitting; Multiple Sclerosis (MS) Primary Progressive; MS (Multiple Sclerosis); MS; Multiple Sclerosis (MS) Secondary Progressive
Keywords: multiple sclerosis; MS; digital tool; UCSF
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to validate a novel, cost-effective method for real-world assessment using patient-acquired "selfie" videos in people with multiple sclerosis. The investigators aim to prove the feasibility and validity of monitoring walking changes remotely through a truly patient-centered, low-burden, low-cost approach. The main question this study aims to answer is: do remotely collected walking and speech videos from a mobile phone match the information investigators can gather from an in person visit?

Participants will collect 5 "selfie" videos at baseline, 3 months, 6 months and 12 months (about 15 minutes every 3 months). They will also come in person at baseline, 6 months, and 12 months for in person data collection (about 1 hour per in person visit).

DETAILED DESCRIPTION:
The investigators aim to validate a novel, cost-effective method for real-world assessment using patient-acquired "selfie" videos. The investigator's preliminary data demonstrate feasibility, validity and utility of this technology, which overcomes limitations of existing digital biomarkers and offers a truly patient-centered, low-burden approach to monitoring and treating diverse people with MS (PwMS). The investigators want to understand the barriers and facilitators to adoption of this approach, as well as the real-world validity and impact of the data generated. This will allow investigators to share the most accessible, generalizable and useful protocols and metrics with the MS community.

This approach to digital tool development prioritizes patients and clinicians. Indeed, the investigators leverage a tool used every day by the general population ("selfie" videos) that recapitulates clinicians' primary examination tool: observing how patients talk and walk.

This approach uses the patient's own device (device agnostic: including smartphones sold after 2010, as well as tablets, laptops or desktops with camera capture), without requiring proprietary software or technology, to collect "selfie" videos - which are ubiquitous in modern life - and provides a link to a secure web portal for simple uploading. The task minimizes burden: it is brief (5 <1min videos), can be done in individuals' own homes, requires no direct or indirect costs, and therefore is accessible to many diverse patients.

Digital biomarkers must demonstrate VALIDITY: sensitivity to subtle change over time, but also relevance to an individual's daily life and function (i.e. veridicality and verisimilitude). Patient selfie videos capture activities relevant in daily life (buttoning a shirt, walking down a hallway, talking about one's morning), across all levels of disability, using assessments that are holistic and that have veridicality and verisimilitude. Furthermore, the metrics show greater sensitivity to change than standard assessments.

Overall objective: Validate video "selfies" as a patient-centered, valid, comprehensive longitudinal data collection method in MS. This approach will be deemed successful if the investigators achieve key metrics informed by implementation science and digital monitoring biomarker validation as necessary for dissemination, which surpass the feasibility, usability or validity of most digital tools currently available for monitoring in MS.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with MS who is above the age of 18 yrs. Participants who are unable to consent for themselves must have a surrogate decision maker or LAR.
* Age > 18 yrs, EDSS - <6.5, own a video recording device (smartphone, tablet, camera etc).

Exclusion Criteria:

* Patient unwilling to participate in the study. Participants unable to consent for themselves who do not have a surrogate decision maker or LAR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A diverse population of adults with MS
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Validate key metrics derived from video "selfies" against the MS Functional Composite (MSFC) | 1 year
  The investigators will optimize key metrics until they show at least 0.75 correlation coefficient with MSFC z scores, as well as individual domains (walking speed/Timed 25 foot walk, processing speed/Symbol digit modalities test, dexterity/9 hole peg test).

SECONDARY OUTCOMES:
Video acquisition protocol usability | 1 year
  The investigators will explore barriers and facilitators to adoption, and iteratively optimize outreach, instructions, video prompts, camera angles and uploading parameters so diverse PwMS can participate in research and care.
Refine single-domain and composite video metrics | 1 year
  Aim 2. Refine single-domain and composite video metrics. Machine learning techniques will generate comprehensive single-domain and holistic metrics of patient functioning that: can be observed asynchronously by clinicians, recapitulate MSFC and EDSS, but are more relevant to daily life than standard metrics.
Validate video metrics' sensitivity to subtle changes over time. | 1 year
  Aim 3. Validate video metrics' sensitivity to subtle changes over time. Over 12 months, the investigators will detect subtle worsening in substantially more patients than by existing single domain / global metrics (MSFC, EDSS), informing the tool's utility in measuring PIRA and response to neurorehabilitation, remyelination, and symptom management.

CONTACTS AND LOCATIONS:
Overall Officials: Riley Bove, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nylander A, Sisodia N, Henderson K, Wijangco J, Koshal K, Poole S, Dias M, Linz N, Troger J, Konig A, Hayward-Koennecke H, Pedotti R, Brown E, Halabi C, Staffaroni A, Bove R. From "invisible" to "audible": Features extracted during simple speech tasks classify patient-reported fatigue in multiple sclerosis. Mult Scler. 2025 Feb;31(2):231-241. doi: 10.1177/13524585241303855. Epub 2024 Dec 17. PMID 39690923
- [Background] Gopal A, Torres WO, Winawer I, Poole S, Balan A, Stuart HS, Fritz NE, Gelfand JM, Allen DD, Bove R. "Self-care selfies": Patient-uploaded videos capture meaningful changes in dexterity over 6 months. Ann Clin Transl Neurol. 2023 Dec;10(12):2394-2406. doi: 10.1002/acn3.51928. Epub 2023 Oct 25. PMID 37877622